CLINICAL TRIAL: NCT02740101
Title: The Role of Oxytocin in Modulating the Effects of Social Feedback on Achieving Personal Goals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-14
Record Dates: First submitted 2016-03-21; First posted 2016-04-15 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: oxytocin; social reward; social punishment

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- oxytocin nasal spray (Experimental): subjects administrating oxytocin were divided into experimental group
  Interventions: Drug: oxytocin treatment
- placebo nasal spray (Placebo Comparator): subjects administrating placebo were divided into controlled group
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: oxytocin treatment — intranasal administration of oxytocin (40 IU)
  Arms: oxytocin nasal spray
Drug: placebo treatment — intranasal administration of placebo (40 IU)
  Arms: placebo nasal spray

SUMMARY:
To examine potential differential effects of receiving various social feedback on achieving personal goals,and whether oxytocin would modulate these effects.

DETAILED DESCRIPTION:
In the present study, 62 healthy male participants participated in the double-blind, placebo-controlled experiment. Investigators aimed to test the idea that whether oxytocin would modulate subjective responses during receiving various social reward and social punishment about the future outcomes of pursuing personal goals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders.

Exclusion Criteria:

* Taking oral contraceptives;
* No history of head injury and medical or psychiatric illness.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rating of Encouragement after receiving specific social feedback | one hour
  There're 96 different social feedback totally for four goals which were divided into four runs consisting of 24 different feedback separately for each goal video.Therefore,subjects were instructed to complete the encouragement rating after receiving each specific feedback. To measure the rating,the investigators used the 9-point likert scale in which one refers to the minimum encouragement while nine refers to maximum encouragement.

SECONDARY OUTCOMES:
Rating of Likeability after receiving specific social feedback | one hour
  There're 96 social feedback totally for four goals which were divided into four runs consisting of 24 feedback separately for each goal video.Therefore,subjects were instructed to complete the likeability rating after receiving each specific feedback. To measure the rating,the investigators used the 9-point likert scale in which one refers to the minimum likeability while nine refers to maximum likeability.

OTHER OUTCOMES:
Rating of Confidence after receiving a series of social feedback | one hour
  There're 96 social feedback totally for four goals which were divided into four runs consisting of 24 feedback separately for each goal video.Furthermore, these 24 feedback were categorized into three types which include 8 feedback separately.Therefore,subjects were instructed to complete the confidence rating after receiving these 8 feedback together. To measure the rating, the investigators used the 9-point likert scale in which one refers to the minimum confidence while nine refers to maximum confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China